CLINICAL TRIAL: NCT03424967
Title: Statistical Learning as a Predictor of Attention Bias Modification Outcome: a Preliminary Study Among Socially Anxious Patients
Brief Title: Statistical Learning as a Predictor of Attention Bias Modification Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Yair Bar-Haim, Professor, Tel Aviv University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAU-SL
Record Dates: First submitted 2018-02-01; First posted 2018-02-07 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Social Anxiety Disorder
Keywords: attention-bias modification; statistical learning; social anxiety disorder; treatment outcome
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ABM therapy (Experimental): The attention bias modification treatment comprises of six computerized sessions, twice a week, in purpose of modulate biases in attention for threat stimuli.
  Interventions: Behavioral: ABM

INTERVENTIONS:
Behavioral: ABM — Participants are trained with a dot-probe task including angry-neutral faces. In 80% of trials the probe appears in place of the neutral face, and in 20% of trials in place of the angry face.
  Other Names: attention bias modification

SUMMARY:
This study examines whether the ability to extract statistical properties from the environment among treatment-seeking patients with social anxiety disorder can predict therapeutic response to attention bias modification (ABM), namely, reduction in symptoms of social anxiety following ABM therapy.

DETAILED DESCRIPTION:
All participants received 6 sessions of ABM therapy away from threat. At baseline participants also completed a gold standard statistical learning task aimed to assess participants' capacity for the extraction of statistical regularity from the environment. The aim of the study is to determine whether the basic ability to extract rules from the environment at baseline could predict clinical improvement of social anxiety symptoms.

ELIGIBILITY:
Inclusion Criteria:

* a signed consent form
* a primary diagnosis of social anxiety disorder
* an age of 18-65

Exclusion Criteria:

* any history or present diagnosis of psychosis
* high risk for harm to self or others
* concurrent posttraumatic stress disorder, eating disorder, or bipolar disorder
* a diagnosis of a neurological disorder (i.e., epilepsy, brain injury)
* drug or alcohol misuse
* a pharmacological treatment that is not stabilized in the past 3 months
* any concurrent psychotherapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-08-02 (Actual); Primary Completion 2017-06-12 (Actual); Study Completion 2017-06-12 (Actual)

PRIMARY OUTCOMES:
The Liebowitz Social Anxiety Scale (LSAS) - Diagnostic Interview scores | 1-2 weeks after treatment completion
  The Liebowitz Social Anxiety Scale is a clinician-rated inventory consisting of 24 items describing socially relevant situations. Each situation is rated in relation to the past week on two sub-scales ranging 0-3: level of fear and level of avoidance experienced in response to these situations. Item scores are summed to a total score ranging 0-144

SECONDARY OUTCOMES:
The Social Phobia Inventory scores | 1-2 weeks after treatment completion
  The Social Phobia Inventory is a self-reported questionnaire comprised of 17 items on a 5-point scale depicting social worries and problems. Participants rate to what extent these situations have bothered them in the past week. Item scores are summed to a total score ranging 0-68.

CONTACTS AND LOCATIONS:
Overall Officials: Yair Bar-Haim, PhD, Principal Investigator — Tel Aviv University
Locations (1):
- Tel Aviv University, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No